CLINICAL TRIAL: NCT01216501
Title: Comparison of Electrophysiological Effects of Sevoflurane and Isoflurane-based Anesthesia in Children Undergoing RF Ablation or Cryoablation for SVT Treatment. A Randomized Double Blind Study.
Brief Title: Sevoflurane and Isoflurane for RF or Cryo Ablation in Children.
Status: Terminated | Type: Observational
Why Stopped: Recruiting was not as anticipated.
Sponsor: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Ludmyla Kachko, MD, Anesthetic physician, Schneider Children's Medical Center, Israel
Other Study IDs: LK-02/2010
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In children, radiofrequency catheter ablation (RFCA) or cryoablation are highly effective treatments for supraventricular tachycardia treatment. General anesthesia is often required to ensure comfort during the prolonged procedure and to assure immobility in order to facilitate accurate mapping and subsequent ablation of the accessory pathway and/or arrhythmogenic focus. Successful anesthetic management of this patient population requires adequate suppression of sympathetic responses during the procedure while electrophysiological parameters remain unaltered for mapping purposes and subsequent ablation. Although Sevoflurane (SEVO) and Isoflurane (ISO) are two commonly used and evaluated volatile anesthetic agents for ablation procedures, comparison of those agents has not been performed previously not in adults, not in children.

Hypothesis Time required for basic EP intervals, successful induction of SVT and successful RFCA or cryoablation in children will not be different between patients undergoing Sevoflurane or Isoflurane-based anesthesia.

DETAILED DESCRIPTION:
In children, radiofrequency catheter ablation (RFCA) or cryoablation are highly effective treatments for supraventricular tachycardia treatment. General anesthesia is often required to ensure comfort during the prolonged procedure and to assure immobility in order to facilitate accurate mapping and subsequent ablation of the accessory pathway and/or arrhythmogenic focus. Successful anesthetic management of this patient population requires adequate suppression of sympathetic responses during the procedure while electrophysiological parameters remain unaltered for mapping purposes and subsequent ablation. Although Sevoflurane (SEVO) and Isoflurane (ISO) are two commonly used and evaluated volatile anesthetic agents for ablation procedures, comparison of those agents has not been performed previously not in adults, not in children.

Hypothesis Time required for basic EP intervals, successful induction of SVT and successful RFCA or cryoablation in children will not be different between patients undergoing Sevoflurane or Isoflurane-based anesthesia.

Patients The study group will include otherwise 200 lthy patients aged 4 to 18 years, with an ASA physical status I or II, who are scheduled for elective radiofrequency ablation or cryoablation to interrupt abnormal foci and/or accessory pathways at Schneider Children's Medical Center of Israel (SCMCI). Written informed consent will be obtained from the patients (from age 12), parent(s) or legal guardian of all participants. Duration of the study- 2 years.

Inclusion criteria: healthy patients aged 4 to 18 years, with an ASA physical status I or II, who are scheduled for elective radiofrequency ablation or cryoablation to treat SVT.

Exclusion criteria: patients with accompanying cardiac defects or other diseases, suspected Malignant Hyperthermia, contraindication to volatile anesthetics use and patients/ parental refusal.

Anesthesia The investigators will use the standard anesthesia protocol. Routine monitoring includes electrocardiography, noninvasive blood pressure measurement, capnography and pulse oximetry.

The patients are randomly divided into two groups according to the last digit of their 9-digit identification number: patients with an odd number are allocated to Sevoflurane (SEVO group) and patients with an even number are allocated to and Isoflurane (ISO group). Preanesthetic medication consists of midazolam given either orally (0.5 mg/kg up to a maximum of 10 mg) or intravenously (2.0 mg) when intravenous (IV) access is established before induction of anesthesia. Anesthesia is induced either via facemask with Sevoflurane (Abbot Laboratories Ltd., UK) in 66% nitrous oxide and 33% oxygen or IV with Propofol (Diprivan, B Braun, Germany) 2.5 mg/kg. In patients who undergo mask induction intravenous line is established after losing the consciousness, Sevoflurane is discontinued and Propofol (2.5 mg/kg) is administerd IV. Before tracheal intubation the lungs will be preoxigenated with 100% O2. Pancuronium (0.1 mg/kg) and Fentanyl (2-4 µg/kg) will be used to facilitate tracheal intubation. After tracheal intubation, the fresh gas flow will be set to 1 l/min O2 and 1 l/min room air for the remainder of the procedure. Thereafter, anesthesia will be maintained with the assigned study drug (SEVO or ISO) in an oxygen/air 50% mixture. In the ISO group, the Isoflurane will be started with an inspiratory fraction of 1MAC and in the SEVO group the Sevoflurane will be started with an inspiratory fraction of 1MAC adjusted for age. Pancuronium is used as the neuromuscular drug during the intraoperative period, as needed.

After induction of anesthesia, a standard baseline programmed stimulation electrophysiological protocol is performed using transvenous endocardial electrodes that allow calculating the following parameters: right atrial refractory period, atrioventricular node effective refractory period, accessory pathway effective refractory period, and right ventricular effective refractory period. Decremental pacing of the right atrium or ventricle allows determining the shortest cycle length during antegrade and retrograde conduction, which is also called the "Wenckebach cycle length," with a 1:1 conduction over the normal atrioventricular node and accessory pathway. Right atrial or ventricular extrastimulus testing involves pacing at a standard drive cycle length of 200, 400 or 600 ms, followed by an extrastimulus coupled (steps of 20 ms from 600-300 ms and steps of 10 ms less than 300 ms) to every eighth drive beat. Baseline intervals measured during sinus rhythm include intraatrial conduction time (PA interval), and atrial-His interval. During induced reciprocating tachycardia, conduction times of each component of the reentrant circuit is measured and included cycle length and atrial-His, His-ventricular, and ventriculoatrial intervals. All electrophysiological measurements is recorded using a standard digitizing tablet at a paper speed of 100 mm/s. Programmed stimulation is performed using a Mennen stimulator, and data is displayed, recorded, and analyzed using a standard computerized multichannel system. If the clinically suspected SVT will not induced during the baseline protocol, isoproterenol (0.03-0.07 µg • kg- 1 • min-1) will be infused, and the protocol repeated until SVT will be induced. After conclusion of the diagnostic study, ablation of the abnormal substrate(s) will be performed using a commercial radiofrequency generator (ATKAR). If needed, the muscle relaxation will be reestablished using pancuronium 0.05mg/kg to allow the ablation be performed during apnea to avoid respiration-related intrathoracic movement. This approach permits application of radiofrequency energy near vital structures, such as the atrioventricular node, with reduced concern of potentially dangerous catheter dislodgement. The final diagnostic electrophysiological study will be repeated at baseline and with isoproterenol (0.03-0.07 µg • kg- 1 • min- 1). Extubation will be performed after the patient awake. Post procedural care will be provided in the recovery room, and patients will be transferred to a ward when hemodynamically stable, fully conscious and able to protect the airway, without pain and severe nausea or active vomiting.

Time Analyses

The following time intervals will be analyzed:

Onset of SVT time - T1 (start of first diagnostic electrophysiological study until induction of first SVT); Diagnostic electrophysiological study time - T2 (start of first diagnostic electrophysiological study until start of ablation); RFCA/ cryoablation procedure time - T3 (start of first diagnostic electrophysiological study until end of final diagnostic electrophysiological study); Wake-up time - T4 (from end of wound dressing to patient exit from the operating room to the post-anesthesia care unit); Total anesthesia time -T5 (from patient entry to operating room to exit from operating room).

If a patient will enter the laboratory in SVT or if SVT will be induced by initial catheter placement, the "onset of SVT time" is designated "0 min." Additionally, the investigators will compare the antegrade effective refractory period of the accessory pathway (antegrade APERP), ventricular effective refractory period (VERP), atrial effective refractory period (AERP), AH interval, and cycle length of circus movement tachycardia (CMT-CL).

In addition, the investigators will compare the incidence of postoperative nausea and vomiting (PONV) in both groups of patients after the procedure (globally and between the patients, who needed Transesophageal Echocardiography - TEE and not). In the case of PONV, Ondansetron (Zofran) will be ordered in the dose of 0.1mg/kg IV. If the PONV continues after ondansetron administration, the second dose of this drug will be given at the dose of 0.1 mg/kg.

The electrophysiologist, who performs the procedure, the patients and their parents are blinded to randomization status. Time points periods will be recorded by the nurse, blinded to the randomization status. The incidence of PONV will be recorded by the nurse in the post anesthesia care unit (PACU), who is blinded to randomization status.

ELIGIBILITY:
Inclusion Criteria:

healthy patients aged 4 to 18 years, with an ASA physical status I or II, who are scheduled for elective radiofrequency ablation or cryoablation to treat SVT.

Exclusion Criteria:

patients with accompanying cardiac defects or other diseases, suspected Malignant Hyperthermia, contraindication to volatile anesthetics use and patients/ parental refusal.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who are scheduled for elective radiofrequency ablation or cryoablation to interrupt abnormal foci and/or accessory pathways at Schneider Children's Medical Center of Israel (SCMCI).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
No statistic information due to the small amount of participants. | No statistic information due to the small amount of participants.
  No statistic information due to the small amount of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ludmyla Kachko, MD, Principal Investigator — Schneider Medical Cebter of Israel
Locations (1):
- Schneider Medical Center of Israel, Petah Tikva, Israel